CLINICAL TRIAL: NCT02922374
Title: Ulcerative Colitis Endoscopic Index of Severity and Fecal Calprotectin to Predict the Reaction to Corticosteroids of Acute Severe Ulcerative Colitis: A Prospective Observational Study
Brief Title: Ulcerative Colitis Endoscopic Index of Severity and Fecal Calprotectin to Predict the Reaction to Corticosteroids of Acute Severe Ulcerative Colitis
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Jinling Hospital, China (Other)
Responsible Party: Principal Investigator, Jianfeng Gong, Associate professor, Jinling Hospital, China
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ASC-UCEIS-FC
Record Dates: First submitted 2016-09-28; First posted 2016-10-04 (Estimated); Last update posted 2016-10-24 (Estimated); Status verified 2016-10

CONDITIONS: Acute Severe Colitis (ASC)
Keywords: acute severe colitis; corticosteroids; UCEIS; fecal calprotectin
MeSH Terms: interventions — Adrenal Cortex Hormones

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- CS (Experimental): Intravenous steroids were started with methylprednisolone 60 mg/d or hydrocortisone 400 mg/d for 3 days.
  Interventions: Drug: corticosteroids

INTERVENTIONS:
Drug: corticosteroids — Intravenous steroids were started with methylprednisolone 60 mg/d or hydrocortisone 400 mg/d for 3 days.

SUMMARY:
For acute severe colitis (ASC) patients, corticosteroids (CS) was recommended as the first-line treatment in the guideline, but patients have a great risk of requiring colectomy or turning to second-line treatment. This study aim to verify the effectiveness of ulcerative colitis endoscopic index of severity(UCEIS) in predicting the reaction to corticosteroids, and explores the possibility that noninvasive marker fecal calprotectin (FC) could act as an alternative to UCEIS.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with a confirmed diagnosis of ASC according to Truelove and Witt's criteria;
2. Patients were generally able to tolerate the flexible colonoscopy before start of CS treatment;

Exclusion Criteria:

1. Patients with incomplete colonoscopy, inadequate fecal sample;
2. Patients with indeterminate diagnosis of ASC (colorectal cancer, Crohn's disease) according to colonoscopy;
3. Patients with infectious colitis, Clostridium difficile and CMV infection, primary immunodeficiency, recent history of immunosuppressant within 3 months.
4. Patients with bowel resection, intestinal anastomotic, and ileum enterostomy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 117 (Actual)
Dates: Start 2013-01; Primary Completion 2016-06 (Actual); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
stool frequency at day 3 | 3 days
  The response to intravenous steroid therapy was judged at day 3 according to Oxford criteria.
C-reactive protein (CRP) at day 3 | 3 days
  The response to intravenous steroid therapy was judged at day 3 according to Oxford criteria.

SECONDARY OUTCOMES:
ulcerative colitis endoscopic index of severity (UCEIS) before treatment | 3 days
  The UCEIS consists of the following three descriptors and was calculated as a simple sum: vascular pattern (scored 0-2), bleeding (scored 0-3), erosions and ulcers (scored 0-3).
Fecal Calprotectin before treatment | 3 days
  FC was measured strictly with the instruction of the commercial test kits.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Generay Surgery, Jinling hosptal, Medical School of Nanjing University, Nanjing, Jiangsu, China